CLINICAL TRIAL: NCT04571762
Title: Feasibility Trial of Individualized Daily Dose Adaptation for Localized Prostate Cancer by Online MR-guided SBRT
Brief Title: Adaptive MR-guided SBRT for Localized Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iAdapt-Prostate
Record Dates: First submitted 2020-07-09; First posted 2020-10-01 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: SBRT; MR-Linac; Adaptive radiotherapy; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Patients with low-risk, intermediate-risk and low-volume metastatic prostate cancer eligible for stereotactic body radiotherapy will be recruited.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT (a fraction dose adapted to the OAR geometry-of-the-day, 5 fractions) performed on the MR-Linac

SUMMARY:
The purpose of this study is to evaluate a technical feasibility of MR-guided SBRT fraction dose adaptation for low-risk, intermediate-risk and low-volume metastatic prostate cancer. .

DETAILED DESCRIPTION:
Hypofractionated SBRT to 36.25 Gy in 5 fractions (fraction dose 7.25 Gy) for low- and intermediate risk prostate cancer is standard of care. Using higher fraction doses that might be beneficial for disease control is not safe in all patients, unless adaptive treatment is performed. In this clinical trial the feasibility of online MR-guided SBRT fraction dose adaptation (between 7 and 8 Gy) for prostate cancer will be investigated. A fraction dose to the planning target volume (PTV) will be adapted to organs-at-risk (OAR) geometry (position, shape and volume) on online planning MRI scans of the treatment day ("geometry-of-the-day"). Thus the investigators hope to maximize treatment individualization.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before any trial specific procedures;
* Males;
* Histologically confirmed adenocarcinoma of the prostate;
* Low (Grade group 1 [Gleason score ≤6], clinical stage T1-2a N0 M0, and PSA < 10 ng/ml) and intermediate (Grade group 2-3 [Gleason score 7], clinical stage T2b-2c N0 M0, PSA 10-20 ng/ml) risk prostate cancer with indications for SBRT with curative intent;
* Newly diagnosed low-volume metastatic prostate cancer with indications for SBRT, in whom metastatic disease was confirmed on a bone scintigraphic scan and soft-tissue imaging done within 3 months of starting androgen deprivation therapy (ADT);
* IPSS <15;
* Age: ≥ 18 years old;
* Karnofsky performance status ≥70;
* Patients able to tolerate long (approximately 60 minutes) treatment time;
* Patients who are willing and able to comply with scheduled visits, treatment, and other trial procedures.

Exclusion Criteria:

* Previous radical treatment for prostate cancer - either radiation therapy (external or brachytherapy), surgery, TUR-P, cryosurgery, or HIFU;
* Contraindications for MRI, e.g., patients with metal fragments or implanted devices that are not MR compatible such as certain types of pacemakers and aneurysm clips or severe claustrophobia;
* Lack of safe contraception;
* Known or suspected non-compliance, drug or alcohol abuse;
* Inability to follow the procedures of the trial, e.g. due to language problems of the participant;
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of online MR-guided SBRT: Number of fractions | At the treatment end (treatment duration 2 weeks)
  Number of fractions when a new online plan on the new patient geometry was successfully generated and applied according to the dosimetric protocol requirements

SECONDARY OUTCOMES:
Rates of adverse events | weekly during treatment and up to 3 months after the treatment end
  Adverse and severe adverse events measured with Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0)
Quantifying intrafraction motion of the prostate (in mm) and organs-at-risk (in mm) | During each treatment session (treatment duration of 2 weeks)
  Changes in the organ motion (in mm) during a treatment session
Quantifying interfraction motion of the prostate (in mm) and organs-at-risk (in mm) | Before each treatment session (treatment duration of 2 weeks)
  Changes in the organ (the prostate and organs-at-risk [in mm]) motion between treatment sessions
Quality of the adapted treatment plan vs. the initial treatment plan | At the treatment end (treatment duration 2 weeks)
  Comparison of radiation doses delivered to the targets and organs-at-risk with the adapted treatment plan vs. the initial treatment plan
Duration of an online adaptive procedure | Before each treatment session (treatment duration 2 weeks)
  Time needed for adapting a treatment plan

CONTACTS AND LOCATIONS:
Overall Officials: Nocolaus Andratschke, MD, Principal Investigator — University of Zurich

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.